CLINICAL TRIAL: NCT04216849
Title: Clinical Study of Umbilical Cord Mesenchymal Stem Cells in the Treatment of Type 2 Diabetic Nephropathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFSC-2019(CR)-06
Record Dates: First submitted 2019-12-17; First posted 2020-01-03 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes With Renal Manifestations
Keywords: human umbilical cord mesenchymal stem cells; type 2 diabetic nephropathy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The volunteers of the experimental group will be given peripheral intravenously a dose of 1.5*10^6/kg human umbilical cord mesenchymal stem cells at 0,8,16,24,32 week.
  Interventions: Biological: human umbilical cord mesenchymal stem cells
- control group (Placebo Comparator): The control group will be given the same dose of saline containing human albumin.
  Interventions: Other: saline

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells — human umbilical cord mesenchymal stem cells were peripheral intravenous infused to experimental group
  Arms: experimental group
Other: saline — Saline solution containing human serum albumin will be infused to the control group
  Arms: control group

SUMMARY:
The study was a 48-week multicenter, randomized, double-blind, placebo-controlled trial that included 8 weeks of pre-screening and lifestyle education, 32 weeks of treatment, and 16 weeks of follow-up.To observe the efficacy and safety of umbilical cord mesenchymal stem cell infusion in Chinese patients with type 2 diabetic nephropathy who received traditional hypoglycemic therapy.

DETAILED DESCRIPTION:
The study was a 48-week multicenter, randomized, double-blind, placebo-controlled trial that included 8 weeks of pre-screening and lifestyle education, 32 weeks of treatment, and 16 weeks of follow-up.We plan to recruit 54 subjects，which were divided into experimental group and control group. The volunteers of the experimental group will be given peripheral intravenously a dose of 1.5*10^6/kg human umbilical cord mesenchymal stem cell (HUC-MSC) at 0,8,16,24,32 week. The control group will be given the same dose of saline. Then centralization visit was conducted every 8 weeks until the 48th week.The primary end points include estimated glomerular filtration rate and urinary albumin creatinine ratio(UACR). The secondary end points include HbA1C,plasma insulin and C-peptide, and insulin dose.

ELIGIBILITY:
Inclusion Criteria (in brief):

* Type 2 diabetes mellitus
* Diabetes duration≤20 years
* 18.5kg/m^2 ≤ BMI< 30 kg/m^2
* 7.5%≤HbA1C≤10%
* UACR≥30mg/gCr
* eGFR ≥45/milliliter/1.73m^2

Exclusion Criteria (in brief):

* Type 1 diabetes mellitus
* tumor history
* Other causes of chronic kidney disease
* Abnormal liver function

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
UACR | 48weeks after treatment
  urinary albumin creatinine ratio

SECONDARY OUTCOMES:
HbA1c | 48weeks after treatment
  HbA1c
insulin/C peptide | 48weeks after treatment
  serum level of insulin/C peptide
insulin dosage | 48weeks after treatment
  insulin dosage
eGFR | 48weeks after treatment
  estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhongming Liu, MD, Principal Investigator — Shanghai East Hospital, Shanghai Tongji University
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China